CLINICAL TRIAL: NCT04687124
Title: N-3 Fatty Acid EPA Supplementation in Cancer Patients Receiving Abdominal Radiotherapy - A Randomised Controlled Trial.
Brief Title: EPA Supplementation in Cancer Patients Receiving Abdominal Radiotherapy -
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jens Rikardt Andersen (Other)
Collaborators: Department of Oncology, Rigshospitalet, Blegdamsvej 9, 2100 Copenhagen (Unknown)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Sponsor - Investigator, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-D-2007-0134
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Abdominal Cancer; Radiotherapy; Complications; Weight Loss; Energy Supply; Protein Deficiency
Keywords: Malnutrition; radiotherapy,; oral nutritional supplements; fish-oil
MeSH Terms: conditions — Weight Loss; Protein Deficiency; Malnutrition | interventions — Fish Oils; Nutrition Assessment; Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomization by sealed envelopes. Stratified for location of cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fish oil (Active Comparator): dietary counselling including an oral nutritional supplement (ONS) containing 2.2 g of n-3 fatty acid EPA (Forticare®)
  Interventions: Dietary Supplement: Fish oil
- standard care (Placebo Comparator): The departmental usual procedure with the possibility of requiring of a dietician when needed
  Interventions: Other: standard care

INTERVENTIONS:
Dietary Supplement: Fish oil — Dietary counseling including an oral nutritional supplement (ONS) containing 2.2 g of n-3 fatty acid EPA (Forticare®)
  Other Names: Dietary counseling
  Arms: Fish oil
Other: standard care — No specified intervention
  Arms: standard care

SUMMARY:
Malnutrition occurs frequently in patients with cancer during and after radiotherapy to the gastrointestinal (GI) area and can lead to negative outcomes. N-3 fatty acids from fish, especially eicosapentaenoic acid (EPA) may possess anticachectic properties. The aim of this study is to investigate the effect of two nutritional interventions; dietary counselling and an oral nutritional supplement (ONS) containing 2.2 g of the n-3 fatty acid EPA (Forticare®) or standard care, including dietary counselling and protein supplementation when needed.

DETAILED DESCRIPTION:
Methods: Outpatients commencing radiotherapy to the GI area due to dissiminated cancer are randomized to receive dietary counselling and daily fish-oil supplementation over a 5-7 week period, or standard care. Outcome parameters are measured at baseline (onset of radiotherapy), week 5, and 12 weeks after commencing radiotherapy, with one additional measurement of body weight at week 2. Quality of life (QoL) is measured using the EORTC QLQ-C30 questionnaire. Radiotherapy-related side effects are assessed using a questionnaire developed specifically for this study. Data from a historical control group collected in a previous observational study is included in this study to compare incidence of weight loss.

ELIGIBILITY:
Inclusion Criteria:

* referred to radiotherapy for dissminated, abdominal cancer
* > 18 years of age
* able to understand and comply with the intervention
* willingness to participate after oral and written conscent

Exclusion Criteria:

* conditions precluding evaluations of end-points
* dementia
* operations planned in the observation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Change in weight (%) | 6 weeks
  accumulated weight-loss or gain in per cent of the weight measured between baseline, end of treatment and at follow-up

SECONDARY OUTCOMES:
energy intake (kJ/day) in % of estimated needs | 6 weeks
  Mean of 3 meausrements in the obeservation period
protein intake (g/kg body weight/day) in % of estimated needs | 6 weeks
  Mean of 3 meausrements in the obeservation period
Quality of life score (EORTC QLQ-C30 version 3.0) points | 6 weeks
  difference - before and after intervention
treatment-related side-effects (VAS) scale | 6 weeks
  questionaire before and after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patursson P, Moller G, Muhic A, Andersen JR. N-3 fatty acid EPA supplementation in cancer patients receiving abdominal radiotherapy - A randomised controlled trial. Clin Nutr ESPEN. 2021 Jun;43:130-136. doi: 10.1016/j.clnesp.2021.03.001. Epub 2021 Mar 16. PMID 34024504